CLINICAL TRIAL: NCT02450006
Title: INtermountain Healthcare Biological Samples Collection Project and Investigational REgistry for the On-going Study of Disease Origin, Progression and Treatment (Intermountain INSPIRE Registry)
Brief Title: Intermountain INSPIRE Registry
Status: Recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1024811
Record Dates: First submitted 2015-04-20; First posted 2015-05-21 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Condition
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Examples of the biological samples that may be collected are as follows (but not limited to):
  * Blood/Plasma
  * Bone Marrow
  * Buccal smear (cheek)
  * Cartilage
  * Cerebrospinal fluid
  * Mucus
  * Saliva
  * Sputum
  * Stool
  * Sweat
  * Synovial fluid
  * Tears
  * Tissue samples (e.g. muscle, skin, nails, tumor, etc)
  * Urine
  * Seminal fluid
  * Genetic material extracted from any biological sample
  * Other biological samples as identified by the Principal Investigator or Co-Investigators and agreed by the patient.
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect biological samples, clinical information and laboratory data from patients diagnosed with any healthcare-related conditions who are seen at facilities affiliated with Intermountain Healthcare, including patients and their family members, and to collect the same information and samples from a general population including disease-free subjects.

DETAILED DESCRIPTION:
This is an observational, non-randomized, open, long-term project to collect a variety of biological samples, in addition to usual or specialized care clinical information and laboratory test results, from patients who present to Intermountain Healthcare-affiliated facilities, with symptoms of any healthcare-related conditions, as well as from a general population including disease-free subjects. The INSPIRE Registry will include all subjects enrolled in the HHD registry (IRB # 1007406, approval date 01- 16-2009) and the cathlab database registry (IRB # 1008366, approval date 10/04/2000), as of IRB approval date of this INSPIRE amended protocol.

Since this is a registry database project, there are no investigational treatments, drugs or procedures associated with participation. Information obtained from this registry project will not have direct or immediate benefit for any of the participants.

Biological samples and subject information will be obtained during diagnostic procedures and/or treatment that are generally part of usual or specialized care for the underlying healthcare-related condition. Sample testing and registry data utilization for various research projects can be initiated only after the appropriate approval is obtained from a registry oversight/management committee, and when appropriate, the Institutional Review Board.

After informed consent is obtained from the patient, the biological samples will be obtained in one of the following ways:

1. During a procedure from access lines inserted for the procedure, or
2. When other ordered lab work is done, or
3. As a separate sample collection if no other lab work is planned. Biological sample collection from the general population may be a separate blood draw and/or sample collection. Participating patients may be asked to provide one or more collections of biological samples. Biological samples may be used in current and future research tests multiple times, or until the sample is consumed. In addition, participating subjects may be asked to complete the IRBreviewed questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any age, any ethnicity, diagnosed with any healthcare-related conditions, presenting to an Intermountain Healthcare-affiliated facility or males or females of any age, any ethnicity, with or without any healthcare-related conditions, including disease-free subjects, from a general population that may include unaffected family members
* Patient or patient's representative has the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures, using a form that is approved by the applicable IRB.

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally-acceptable representative to provide informed consent for any reason.
* Other conditions that in the opinion of the Principal Investigator or Co-Investigator(s) may increase risk to the subject and/or compromise the quality of the registry project.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with any healthcare-related conditions who are seen at facilities affiliated with Intermountain Healthcare, including patients and their family members, the general population, including disease-free subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2015-04; Primary Completion 2050-04 (Estimated); Study Completion 2050-04 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center and Intermountain Clinics, Murray, Utah, United States

REFERENCES:
- [Derived] Horne BD, May HT, Muhlestein JB, Le VT, Bair TL, Knowlton KU, Anderson JL. Association of periodic fasting with lower severity of COVID-19 outcomes in the SARS-CoV-2 prevaccine era: an observational cohort from the INSPIRE registry. BMJ Nutr Prev Health. 2022 Jul 1;5(2):145-153. doi: 10.1136/bmjnph-2022-000462. eCollection 2022 Dec. PMID 36619318
- [Derived] Bartholomew CL, Muhlestein JB, Anderson JL, May HT, Knowlton KU, Bair TL, Le VT, Bailey BW, Horne BD. Association of periodic fasting lifestyles with survival and incident major adverse cardiovascular events in patients undergoing cardiac catheterization. Eur J Prev Cardiol. 2022 Jan 11;28(16):1774-1781. doi: 10.1093/eurjpc/zwaa050. PMID 33624026